CLINICAL TRIAL: NCT03682900
Title: Expanding the Click City Tobacco Prevention Program to Include E-cigarettes and Other Novel Tobacco Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Behavioral Intervention Strategies, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DA044025; 2R44DA044025 (NIH); NCT05730322 (obsolete NCT alias)
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Results first posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Tobacco Use
Keywords: e-cigarettes; prevention; middle school; smoking
MeSH Terms: conditions — Tobacco Use; Vaping; Smoking

STUDY DESIGN:
Intervention Model Description: Schools were stratified by state, size of school (small, medium, large) and desired start date and randomized to intervention or control. Intervention and control schools were yoked for the timing of assessments (baseline and follow-up assessments).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Click City Tobacco Prevention Program (Experimental): Participation consisted of a baseline assessment one-week prior to starting the program, and a follow-up assessment one-week following completion of the program. The expectation was that students complete two lessons a week of the computer-based program over a four-week period.
  Interventions: Other: Click City®: Tobacco
- Control: Usual Tobacco Prevention Curriculum (Experimental): Students in control schools completed the baseline and follow-up assessments during the same week as students in their yoked intervention school. The expectation was that students would participate in the standard tobacco curriculum over this period.
  Interventions: Other: Usual Tobacco Curriculum

INTERVENTIONS:
Other: Click City®: Tobacco — A computer-based program assigned to students designed to prevent subsequent tobacco use. Students complete one 15 to 20 minute lesson two times a week for four weeks.
  Arms: Intervention: Click City Tobacco Prevention Program
Other: Usual Tobacco Curriculum — Students complete their usual curriculum designed to prevent tobacco use.
  Arms: Control: Usual Tobacco Prevention Curriculum

SUMMARY:
The goal of this study is to modify a smoking prevention program for 5th and 6th grade students to also target vaping e-cigarettes. Aims were to modify the program along with associated materials and to conduct a trial with 5th grade students in the school setting to see how well the updated program worked. Students either participated in the four-week computer based program or continued with their usual tobacco prevention curriculum.

This study showed that students who received the computer program reduced their intentions and willingness to use e-cigarettes or smoke in the future more than did students who used their usual tobacco curriculum.

DETAILED DESCRIPTION:
Given the increase in prevalence of e-cigarette use among youth, investigators modified a smoking prevention program to not only target smoking but also vaping e-cigarettes. Investigators conducted a pragmatic randomized trial with 5th grade students in schools across Arizona and Oregon to evaluate the effectiveness of the updated program in a "real-world" setting. Forty-five schools were randomized to the intervention condition, wherein students used the updated version of Click City®: Tobacco, or the control condition, wherein students were taught their usual tobacco prevention curriculum. Students in the intervention schools decreased their intentions and willingness to use e-cigarettes and cigarettes significantly, as compared to students in control schools. The intervention also significantly changed all etiological mechanisms. The effects on all outcomes of the intervention were similar as a function of state (Arizona vs Oregon), gender, ethnicity (Hispanic vs not Hispanic), and historical timing (prior to school closures in 2020 vs after schools re-opened in 2022). The intervention was also more effective for at-risk students, as defined by student's previous tobacco use, current family use and/or high in sensation seeking. Close to 90% of the students completed the entire program, and most completed it in 3 to 4 weeks, the expected time frame. The effectiveness of the updated Click City®: Tobacco was demonstrated in a "real world" setting and findings suggested that all students can potentially benefit from the program.

ELIGIBILITY:
Inclusion Criteria:

* A 5th grade student in one of the recruited schools
* Student speaks English as a first or second language
* Passive parental consent to participate

Exclusion Criteria:

* Special needs students identified by the classroom teacher as a student who would not understand the questionnaire or the program
* Teacher indicates that they cannot comprehend English.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2673 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judy A Andrews, PhD, Principal Investigator — Oregon Research Behavioral Intervention Strategies, Inc.; Judith S. Gordon, PhD, Principal Investigator — University of Arizon
Locations (1):
- Oregon Research Behavioral Intervention Strategies, Inc., Springfield, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study took place in the schools from January 6, 2020 through June 10, 2022. Within 43 recruited schools, 2906 5th grade students were initially eligible for participation. Among these students, 111 had parents who actively declined their participation, resulting in 2795 students within randomized schools, as eligible for enrollment. Among these, 2673 were enrolled in the study, as defined by completing the baseline and/or follow-up assessment.
Pre-assignment Details: No events.
Units Other Than Participants: schools
Groups:
- Intervention: Students in intervention schools were expected to complete Click City®: Tobacco, a computer-based program designed to prevent subsequent tobacco use. Students were expected to do a 15 to 20 minute lesson two times a week for four weeks. Participation also consisted of a baseline assessment one-week prior to starting the program, and a follow-up assessment one-week following completion of the program.
- Control: Students in control schools were expected to complete their usual tobacco curriculum, designed to prevent tobacco use. Students completed the baseline and follow-up assessments during the same week as students in their yoked intervention school. The expectation was that students would participate in the standard tobacco curriculum over the same period that students in the intervention group completed Click City®: Tobacco.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 1346; 22 schools | 1327; 21 schools
Completed | 1346; 22 schools (Students completed either the baseline assessment or the follow-up assessment to be considered enrolled in the study and in the final sample.) | 1327; 21 schools
Not Completed | 0; 0 schools | 0; 0 schools

BASELINE CHARACTERISTICS:
Population: The baseline analyses are based on those who completed the baseline assessment. Students enrolled in the study completed either the baseline assessment, the follow-up assessment or both assessments.
Groups:
- Intervention: Students in the intervention group were expected to complete Click City®: Tobacco, a computer-based program designed to prevent subsequent tobacco use. Students were expected to do a 15 to 20 minute lesson two times a week for four weeks. Participation also consisted of a baseline assessment one-week prior to starting the program, and a follow-up assessment one-week following completion of the program.
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 1233 | 1215 | 2448
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1233 | 1215 | 2448
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: boy | 576 | 545 | 1121
  Gender: girl | 594 | 580 | 1174
  Gender: neither boy nor girl | 59 | 44 | 103
  Gender: not reported (missing) | 4 | 46 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 370 | 371 | 741
  Not Hispanic or Latino | 863 | 840 | 1703
  Unknown or Not Reported | 0 | 4 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 16 | 19 | 35
  Asian | 29 | 23 | 52
  Native Hawaiian or Other Pacific Islander | 6 | 2 | 8
  Black or African American | 29 | 44 | 73
  White | 1093 | 1067 | 2160
  More than one race | 60 | 56 | 116
  Unknown or Not Reported | 0 | 4 | 4
Student's use of tobacco prior to the trial [Count of Participants; unit: Participants]
  Students used tobacco | 82 | 122 | 204
  Students did not use tobacco | 1145 | 1091 | 2236
  Not reported | 6 | 2 | 8
Family members' current use of tobacco [Count of Participants; unit: Participants] — This variable was assessed by four items: (a) "Do any of your brothers, sisters, stepbrothers or stepsisters smoke cigarettes?"; (b) ". . . vape e-cigarettes?"; (c) Does your mom/stepmother smoke or father/step-father smoke cigarettes?"; (d) . . . "vape e-cigarettes?". If the student answered in the affirmative to any of the four items, they were considered to be a member of an nicotine-using family
  Participants
    Family member uses nicotine | 489 | 523 | 1012
    Family member does not use nicotine | 741 | 689 | 1430
    Not reported | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Behavioral Intentions to Vape E-cigarettes
Description: Measured by two items, assessing the student's intentions regarding vaping e-cigarettes as a teen or as a grown-up. Responses were on a five-point scale ranging from "definitely not" (1) to "definitely will" (5). The scale was created by summing the two items with potential range from 2 to 10. A higher score means a worse outcome.
Time Frame: baseline; six months
Population: Students are nested within schools. Although schools are the unit of randomization, students are the unit of analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention: Participation consisted of a baseline assessment one-week prior to starting the program, and a follow-up assessment one-week following completion of the program. The expectation was that students complete two lessons a week of the computer-based program over a four-week period.
  Click City®: Tobacco: A computer-based program assigned to students designed to prevent subsequent tobacco use. Students complete one 15 to 20 minute lesson two times a week for four weeks.
- Control: Students in control schools completed the baseline and follow-up assessments during the same week as students in their yoked intervention school. The expectation was that students would participate in the standard tobacco curriculum over this period.
  Usual tobacco curriculum: Students complete their usual curriculum designed to prevent tobacco use
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1346 | 1327
score on a scale | -.14 (1.325) | 0.0 (1.20)
Statistical Analysis 1: Comparison: Intervention vs Control; Data were analyzed using a general linear mixed model with students nested within schools and schools nested within condition; Test type: Superiority; p = .000, Mixed Models Analysis — A one tailed test was used, as the intervention is expected to be superior than the control group. The criterion for significance was p <. 05; There were no adjustments made for multiple comparisons

2. Primary Outcome: Change in Behavioral Intentions to Smoke Cigarettes
Description: Measured by two items assessing the student's intentions to smoke cigarettes as a teen or as a grown-up. Responses were on a five-point scale ranging from "definitely not" (1) to "definitely will" (5). The scale was created by summing the two items with a potential range from 2 to 10. A higher score means a worse outcome.
Time Frame: baseline; six weeks
Population: Students are nested within schools. Although schools are the unit of randomization, students are the unit of analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1346 | 1327
score on a scale | -.12 (1.026) | .04 (1.125)
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .000, Mixed Models Analysis — The a prior threshold for statistical significance is set at p<.05; one tailed test, as the intervention is expected to be superior than the control group. The p-value is not adjusted for multiple comparisons

3. Primary Outcome: Change in Willingness to Vape E-cigarettes
Description: Measured by four items, assessing the student's willingness to vape e-cigarettes if the opportunity presented itself (with a group of kids with e-cigaretes available and with kids who are vaping and you want to be a part of the group. Willingness to vape was assessed for two levels, "try a few vapes" and "try vaping several times in a row". Responses were on a five point scale, "not at all willing" (1) to "very willing" (5) and were summed for the two scenarios and two levels, yielding a scale from 4 to 20. A higher score means a worse outcome.
Time Frame: baseline; six weeks
Population: Students are nested within schools. Although schools are the unit of randomization, students are the unit of analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1346 | 1327
score on a scale | -.07 (1.77) | .14 (2.00)
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .044, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]

4. Primary Outcome: Change in Willingness to Smoke Cigarettes
Description: Measured by four items, assessing the student's willingness to smoke cigarettes if the opportunity presented itself ("with a group of kids with cigarettes available" and "with kids who are smoking and you want to be a part of the group". Willingness to smoke was assessed for two levels, "try a few puffs" and "smoking the whole cigarette". Responses were on a five point scale, "not at all willing" (1) to "very willing" (5) and were summed for the two scenarios and two levels, yielding a scale from 4 to 20. A higher score means a worse outcome.
Time Frame: baseline; six weeks
Population: Students were nested within schools. Students are the unit of analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1346 | 1327
score on a scale | -.05 (1.42) | .12 (1.635)
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .033, Mixed Models Analysis — The p-value is not adjusted for multiple comparisons. The a priori threshold for significance is p<.05

5. Secondary Outcome: Change in Favorable Social Images of Smokers
Description: Students rate what they "think kids who smoke are like" using a three-point rating scale from "not at all like this" (1) to "very much like this" (3) to rate three attributes, "popular", "cool or neat" and "exciting". The three attributes are summed and the potential score goes from 3 to 9. A higher score means a worse outcome.
Time Frame: baseline; six weeks
Population: Students are nested within schools. Schools were randomly assigned to an arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1346 | 1327
score on a scale | -.87 (1.175) | -.16 (1.53)
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .001, Mixed Models Analysis — All probabilities for secondary outcomes were listed as p = .000 within the analysis program. A p value of < .05 is considered significant. All statistical tests are one-tailed. The p-value is not adjusted for multiple comparisons

6. Secondary Outcome: Change in Favorable Social Images of E-cigarette Vapers
Description: Students rate what they "think kids who vape e-carettes are like" using a three-point rating scale using "not at all like this" (1) to "very much like this" (3) to rate three attributes, "popular", "cool or neat" and "exciting". The three attributes are summed and the potential score ranges from 3 to 9. A higher score means a worse outcome.
Time Frame: baseline; six weeks
Population: Students are nested within schools and schools are randomly assigned to condition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1346 | 1327
score on a scale | -.87 (1.255) | -.17 (1.635)
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

7. Secondary Outcome: Change in Normative Social Images of Smokers
Description: Students rate what they "think other 5th grade kids think kids who smoke cigarettes are like" using a three-point rating scale using "not at all like this" (1) to "very much like this" (3) to rate three attributes, "popular", "cool or neat" and "exciting". The three attributes are summed and the potential score ranges from 3 to 9. A higher score means a worse outcome.
Time Frame: baseline; six weeks
Population: Students are nested within schools. Although schools are the unit of randomization, students are the unit of analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1327 | 1346
score on a scale | -.56 (1.015) | -.16 (1.315)
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

8. Secondary Outcome: Change in Normative Social Images of Vapers
Description: Students rate what they "think other 5th grade kids think kids who vape e-cigarettes are like" using a three-point rating scale using "not at all like this" (1) to "very much like this" (3) to rate three attributes, "popular", "cool or neat" and "exciting". The three attributes are summed and the potential score ranges from 3 to 9. A higher score means a worse outcome.
Time Frame: baseline; six weeks
Population: Students are nested within schools. Although schools are the unit of randomization, students are the unit of analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1346 | 1327
score on a scale | -.62 (1.08) | -.19 (1.445)
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]

9. Secondary Outcome: Change in Perception of Friends Approval of Smoking
Description: Students indicated their perception of friends' approval of their smoking of each of three levels of cigarettes, trying, smoking a few, and smoking a few a day. Responses to each item ranged from "yes" (1) to "no" (3). Summing the three levels ranged from 3 to 9, with a higher score means a better outcome.
Time Frame: baseline; six weeks
Population: Students are nested within schools. Although schools are the unit of randomization, students are the unit of analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1346 | 1327
score on a scale | -.10 (.78) | .01 (.92)
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

10. Secondary Outcome: Change in Perception of Friends Approval of Vaping
Description: Students indicated their perception of friends' approval of their vaping of each of three levels of cigarettes, trying, vaping a few, and vaping a few a day. Responses to each item ranged from "yes" (1) to "no" (3). Summing the three levels ranged from 3 to 9, with a higher score indicating a better outcome.
Time Frame: baseline; six weeks
Population: Students nested within schools.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1346 | 1327
score on a scale | -.14 (.93) | .04 (1.11)
Statistical Analysis 1: Comparison: Intervention vs Control; Data were anlyzed using a general linear mixed model with students nested within schools and schools nested within condition; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

11. Secondary Outcome: Change in Perception of Risk of Second-hand Smoke Exposure
Description: Perception of the risk of getting four diseases ("breathing problems", "asthma", "ear infections" "heart disease", and "lung disease or cancer") as a result of being "often around someone who smokes". Responses for each disease are on a five point scale ranging from "no chance" (1) to "certain to happen" (5). Items were summed to form a scale. The total scale of five items ranged from 4 to 20. A higher score means a better outcome.
Time Frame: baseline; six weeks
Population: Students are nested within schools. Although schools are the unit of randomization, students are the unit of analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1346 | 1327
score on a scale | 3.00 (4.05) | .90 (3.905)
Statistical Analysis 1: Comparison: Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

12. Secondary Outcome: Change in Perception of Risk of Second-hand Vape Exposure
Description: Perception of the risk of getting each of four diseases ("breathing problems", "asthma", "ear infections" , and "lung disease or cancer") as a result of being "often around someone who vapes". Responses for each disease are on a five point scale ranging from "no chance" (1) to "certain to happen" (5). Items were summed to form a scale. The total scale of four items ranged from 4 to 20. The follow-up measure was subtracted from the baseline measure, with a higher score indicating a favorable outcome.
Time Frame: baseline; six weeks
Population: Students are nested within schools. Although the school was the unit of randomization, the student is the unit of analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1346 | 1327
score on a scale | 3.27 (4.195) | 1.02 (3.955)
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

13. Secondary Outcome: Change in Perception of Risk of Cumulative Consequences of Smoking
Description: Perception of risk of getting three diseases (lung cancer, serious breathing diseases, and heart disease) as a result of three levels of cigarettes, "one", "a few cigarettes a day for two years", "a pack of cigarettes a day for two years". Responses for each disease and each level ranged from "no chance" (1) to "certain to happen" (5). Items were summed to form a scale. The total scale of nine items ranged from 9 to 45. A higher score means a better outcome.
Time Frame: baseline; six weeks
Population: Students are nested within schools. Students are the unit of analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1346 | 1327
score on a scale | 1.60 (8.365) | -.09 (8.38)
Statistical Analysis 1: Comparison: Intervention vs Control; Data were analyzed using a gneral linear mixed model with students nested within schools and schools nested within condition; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

14. Secondary Outcome: Change in Perception of Risk of Cumulative Consequences of Vaping
Description: Perception of risk of getting three diseases (lung cancer, serious breathing diseases, and heart disease) as a result of three levels of e-cigarettes, "one time", "a few times a day for two years", "Twenty or more times a day for two years'. Responses for each disease and each level ranged from "no chance" (1) to "certain to happen" (5). Items were summed to form a scale. The total scale of nine items ranged from 9 to 45. A higher score means a better outcome.
Time Frame: baseline; six weeks
Population: Students are nested with schools, which are randomized to condition. Students are the unit of analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1346 | 1327
score on a scale | 3.05 (8.410) | .35 (8.335)
Statistical Analysis 1: Comparison: Intervention vs Control; Data were anlayzed using a general linear mixed model with students nested within schools and schools within condition; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

15. Secondary Outcome: Change in Perception of Risk of Smoking Each Cigarette
Description: Risk of smoking each cigarette was measured by two items indicating what would happen to a 12 year old who started smoking, "every cigarette smoked hurts them a bit" and "The very next cigarette probably won't hurt their bodies". The response scale was a five-point scale ranging from "strongly agree" (1) to "strongly disagree" (5). The scale consisted of summing both items with the former item reversed scored. Scale scores ranged from 2 to 10. A higher score indicated a more favorable outcome.
Time Frame: baseline; six weeks
Population: Students are nested within schools. Although schools are the unit of randomization, students are the unit of analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1346 | 1327
score on a scale | .68 (1.650) | .19 (1.665)
Statistical Analysis 1: Comparison: Intervention vs Control; Data were analyzed uisng a general linear mixed model with students nested within schools and schools nested within condition; Test type: Superiority; p < .001, Mixed Models Analysis — All probabilities for secondary outcomes were listed as p = .000 within the analysis program. Apriori, a p value of < .05 is considered significant. All statistical tests are one-tailed. The p-value is not adjusted for multiple comparisons

16. Secondary Outcome: Change in Perception of Risk of Vaping Each E-cigarette
Description: Risk of vaping each e-cigarette was measured by two items indicating what would happen to a 12 year old who started vaping, "every e-cigarette vaped hurts them a bit" and "the very next e-cigarette probably won't hurt their bodies". The response scale was a five-point scale ranging from "strongly agree" (1) to "strongly disagree" (5). The scale consisted of summing both items with the former item reversed scored. Scale scores ranged from 2 to 10. A higher score indicated a more better outcome.
Time Frame: baseline; six weeks
Population: Students are nested within schools. Schools are the unit of assignment while students are the unit of analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1346 | 1327
score on a scale | .78 (1.685) | .24 (1.725)
Statistical Analysis 1: Comparison: Intervention vs Control; Data were analyzed using a general linear model with students nested within schools and schools nested within condition; Test type: Superiority; p < .001, Mixed Models Analysis — All probabilities for secondary outcomes were listed as p = .000 within the analysis program. A p value of < .05 is a priori considered significant. All statistical tests are one-tailed. The p-value is not adjusted for multiple comparisons

17. Secondary Outcome: Change in Perception of Risk of Addiction From Smoking
Description: Change in perception of risk of getting addicted to smoking as a result of five levels of smoking, ranging from "one time" to a "a pack of cigarettes a day for five years". Responses for each level were on a five-point scale ranging from "no chance" (1) to "certain to happen" (5). Items were summed to form a scale. The total scale of the five items ranged from 5 to 25. A higher score means a better outcome.
Time Frame: baseline; six weeks
Population: Students are nested within schools. Although schools are the unit of randomization, students are the unit of analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1346 | 1327
score on a scale | 2.27 (5.905) | .72 (6.045)
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

18. Secondary Outcome: Change in Perception of Risk of Addiction From Vaping
Description: Perception of risk of getting addicted to vaping as a result of vaping five levels of increasing quantities of e-cigarettes, ranging from "one time" to a "20 times a day for 5 years". Responses for each level were on a five-point scale ranging from "no chance" (1) to "certain to happen" (5). Items were summed to form a scale. The total scale ranged from 5 to 25. A higher score means a better outcome.
Time Frame: baseline; six weeks
Population: Students are nested within schools. Although schools are the unit of randomization, students are the unit of analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1346 | 1327
score on a scale | 2.49 (5.92) | .73 (5.98)
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

19. Secondary Outcome: Change in Perception of Control Over Quitting Smoking
Description: Students answered "how much control do you think you would have over quitting smoking" using a four-point response scale ranging from "no control" (1) to "total control" (4). Perception of control was indicated within four levels of increasing quantities of cigarettes, ranging from "tried a cigarette" to "a pack a day for five years". The four Items were summed to form a scale with the total scale ranging from 4 to 16. A higher score means a worse outcome.
Time Frame: baseline; six weeks
Population: Students are nested within schools. Although schools are the unit of randomization, students are the unit of analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1346 | 1327
score on a scale | -8.53 (13.265) | -1.90 (14.605)
Statistical Analysis 1: Comparison: Intervention vs Control; Data were anlyzed using a general linear model mixed model with students nested within schools and schools nested within condition; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

20. Secondary Outcome: Change in Perception of Control Over Vaping
Description: Students answered "how much control do you think you would have over quitting vaping e-cigarettes" using a four-point response scale ranging from "no control" (1) to "total control" (4). Students indicated thier perception of control within each of four levels of increasing quantities of e-cigarettes, ranging from "tried vaping" to "20 times a day for five years". The four Items were summed to form a scale with the total scale ranging from 4 to 16. A lower score indicated a better outcome.
Time Frame: baseline; six weeks
Population: Students are nested within schools. Although schools are the unit of randomization, students are the unit of analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1346 | 1327
score on a scale | -7.93 (13.60) | -1.99 (14.78)
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

21. Secondary Outcome: Change in Perception of Risk of Difficulty Quitting Smoking
Description: Perception of risk of difficulty quitting smoking as a result of vaping five levels of increasing quantities of cigarettes smoked, ranging from "one cigarette" to a " a pack of cigarettes a day for 5 years". Responses for each level were on a five-point scale ranging from "Very easy" (1) to "Very difficult" (5). Items were summed to form a scale. The total scale ranged from 5 to 25. A higher score meant a better outcome.
Time Frame: baseline; six weeks
Population: Students are nested within schools. Although schools are the unit of randomization, students are the unit of analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1346 | 1327
score on a scale | 2.39 (4.485) | .19 (4.865)
Statistical Analysis 1: Comparison: Intervention vs Control; Data were analyzed using a general linear mixed model with students nested within schols and schools nested within condition; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

22. Secondary Outcome: Change in Perception of Risk of Difficulty Quitting Vaping
Description: Perception of risk of difficulty of quitting vaping as a result of vaping five levels of increasing quantities of e-cigarettes vaped, ranging from "one time" to a " 20 times a day for 5 years". Responses for each level were on a five-point scale ranging from "Very easy" (1) to "Very difficult" (5). Items were summed to form a scale. The total scale ranged from 5 to 25. A higher score means a better outcome.
Time Frame: baseline; six weeks
Population: Students are nested within schools. Although schools are the unit of randomization, students are the unit of analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1346 | 1327
score on a scale | 2.38 (4.645) | .16 (4.970)
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected across the six weeks participation window of each student.
Description: If adverse events are reported, they are referred to a clinical psychologist and evaluated. No adverse events were reported.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/1346 | 0/1327
Serious Adverse Events (participants affected / at risk) | 0/1346 | 0/1327
Other Adverse Events (participants affected / at risk) | 0/1346 | 0/1327

LIMITATIONS AND CAVEATS:
The trial was interrupted half way through by school closures as a result of the pandemic. The trial was re-instated two years later. There were no differences on the effect of the intervention due to timing of the implementation of the trial (prior to versus following school closures). Technical problems led to inability to match IDs. The data for these participants was dropped from that portion of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT03682900/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT03682900/ICF_001.pdf